CLINICAL TRIAL: NCT06992115
Title: Randomized Controlled Trial of MIND Diet for Neuroprotection and Symptom Management in MS
Brief Title: A Study of the MIND Diet for Persons With Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ilana Katz Sand, Associate Professor, Neurology; Associate Director, CGD Center for MS, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 23-0300; RG-2407-43743 (Other Grant/Funding Number: National Multiple Sclerosis Society (NMSS))
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Diet
MeSH Terms: conditions — Multiple Sclerosis | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Neurological exams and functional & cognitive assessments will be conducted by trained staff who are masked from the participant's diet assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIND Diet (Experimental): Participants randomized to the intervention arm will change their dietary patterns to adhere to the MIND diet for one year after randomization.
  Interventions: Behavioral: Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Diet; Behavioral: Small Group
- Continue Diet (Placebo Comparator): Participants randomized to the control arm will continue their current dietary habits, without major changes, for one year after randomization. Participants will not receive diet education in small group.
  Interventions: Behavioral: Small Group

INTERVENTIONS:
Behavioral: Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Diet — A dietary pattern which promotes the intake of olive oil, fish, leafy greens & other vegetables, fruits, whole grains, and legumes, and discourages processed foods, red meat, and sugar.
  Arms: MIND Diet
Behavioral: Small Group — Education and social support on topics related to multiple sclerosis such as disease-modifying therapies and MRI in MS.

SUMMARY:
This study will assess the impact of a MIND (Mediterranean-DASH Intervention for Neurodegenerative Delay) diet on brain health and MS symptoms. Participants will be randomly assigned to one of two arms: the diet intervention arm or the "continue current diet"/control arm. Participants randomized to the dietary intervention arm will change their diet to follow a MIND dietary pattern for one year; diet-related education and programming is provided to support this change. Participants randomized to the continue/control arm will be asked to continue their current dietary habits, without major change for one year; multiple sclerosis (MS) MS-related related education and programming (unrelated to diet) is provided. All participants will be asked to provide blood & stool samples and to complete online questionnaires & three in-person assessments.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the effects of a Mediterranean-style dietary intervention on neuroprotection and symptom management in MS with an early phase II, randomized, controlled clinical trial. Participants will be randomized-stratified by MS phenotype and treatment type-to the diet intervention arm (change current diet to a MIND diet) or the continue/control arm (no major change in current dietary habits).

All patients will participate in a baseline visit, and 6 month visit, a 12 month (end of study visit), and meet with small support groups between study visits.

Participants will also complete online questionnaires, undergo functional & cognitive assessments, and contribute blood & stool samples while on protocol.

The diet intervention arm will receive MIND diet-related education and support from the study dietitian and the principal investigator; virtual small group environments will facilitate discussion about participants' experience and potential challenges with MIND diet adherence and ways to overcome them. Virtual groups will meet weekly for the first month, then monthly through month 12.

The continue current dietary habits /control arm will receive MS-related education and support unrelated to diet from members of the study team and the principal investigator. Group meeting topics and schedules will be provided in advance to offer flexibility; participants are required to attend 6 virtual small group meetings but are invited to join as many as desired.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 years, inclusive
* MS diagnosis, on any treatment (including no treatment)
* MIND diet score of ≤8 at baseline
* NfL parameters determined by age

Exclusion Criteria:

* Diagnosis of an additional neurodegenerative disease (e.g. Alzheimer's) or other serious neurological condition (e.g. stroke)
* Current serious medical condition that could impact the ability to participate or influence study results (e.g. cancer, HIV)
* Pregnancy/planning during study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma neurofilament light chain (NfL) | Baseline, 6-months, and at 12-months
  Plasma NfL quantification will be reported in units of pg/ml.

SECONDARY OUTCOMES:
Neurological Fatigue Index-MS (NFI-MS) | Baseline, 6-months, and at 12-months
  The NFI-MS is a brief (5-10-minute completion time), 23-item survey that measures fatigue in MS. Each question corresponds to a subscale that describes different facets of MS fatigue: physical (range 0-8), cognitive (range 0-4), relief by diurnal sleep or rest (range 0-6), and abnormal nocturnal sleep & sleepiness (range 0-5). A summary score (range 0-30) can be calculated based on the responses from 10 of the items on the questionnaire. Scores are based on the respondent's level of agreement with each statement (0, Strongly Disagree; 1, Disagree; 2, Agree; 3, Strongly Agree); higher scores indicate higher levels of fatigue.
The Expanded Disability Status Scale (EDSS) | Baseline, 6-months, and at 12-months
  The Expanded Disability Status Scale (EDSS) helps to describe the extent to which one's MS affects their everyday functionality based on a neurological and physical exam. Total scale is scored from 1-10, with a higher score indicating greater levels of disability due to MS.
The Symbol-Digit Modalities Test (SDMT) | Baseline, 6-months, and at 12-months
  The Symbol Digit Modalities Test (SDMT) presents a series of nine symbols, each paired with a single digit in a key at the top of a stimulus page. Subjects voice the number associated with each symbol as rapidly as possible. The examiner records the total amount of responses completed. The task continues for 90 seconds with the research staff recording responses. The SDMT score ranges from 0 to 110, with higher values representing a better outcome in cognitive processing speed.
California Verbal Learning Test (CVLT-II) | Baseline, 6-months, and at 12-months
  The California Verbal Learning Test-Second Edition (CVLT-II) is a widely used neuropsychological assessment designed to evaluate verbal learning and memory. It requires individuals to recall words across multiple trials, measuring encoding, recall strategies, and recognition accuracy.
  Scores are based on the number of correctly recalled words across different conditions, including immediate free recall, short-delay free & cued recall, long-delay free & cued recall. Each trial is scored separately, with higher scores (range 0-16) indicating the successful recall of a word; raw scores are converted to a T-score based on age-and-sex-matched normative data.
Brief Visuospatial Memory Test (BVMT-R) | Baseline, 6-months, and at 12-months
  The Brief Visuospatial Memory Test-Revised (BVMT-R) is a neuropsychological assessment designed to measure visuospatial learning and memory. It consists of multiple trials where individuals are asked to recall and recognize geometric figures after a brief exposure.
  Scores are based on the number and accuracy of correctly recalled figures across trials. Each trial is scored separately, with higher scores (range 0-12) indicating the successful recall of a word; raw scores are converted to a T-score and percentile based on age-matched normative data.
  Higher scores (range 0-9) indicating better visuospatial memory performance
The 9-Hole Peg Test (9HPT) | Baseline, 6-months, and at 12-months
  The 9-Hole Peg Test (9HPT) assesses finger dexterity and fine motor coordination. Participants place and remove pegs from a board as quickly as possible, with completion time serving as the primary measure, where faster times indicate better performance.
Timed 25-Foot Walk (T25FW) | Baseline, 6-months, and at 12-months
  Timed 25-Foot Walk (T25FW) evaluates walking speed and ability; a faster completion time on these tests indicates a better performance.
The 2-Minute Walk Test | Baseline, 6-months, and at 12-months
  The 2-Minute Walk Test measures endurance, indicated by a greater distance walked over a two-minute interval.
Multiple Sclerosis Impact Scale (MSIS-29) | Baseline, 6-months, and at 12-months
  The MSIS-29 is a 29-item questionnaire designed to assess the extent to which individuals feel their MS impacts their daily life. Respondents rate the effect of MS on different aspects of their life using a 5-point scale (1 = Not At All, 2 = A Little, 3 = Moderately, 4 = Quite A Bit, 5 = Extremely). The questionnaire includes two subscales: a physical subscale with 20 items and a psychological subscale with 9 items. The total range for each subscale is transformed to a 0-100 scale, with higher scores indicating a greater perceived negative impact of MS.
Multiple Sclerosis Cognitive Scale (MSCS) | Baseline, 6-months, and at 12-months
  The MSCS is an 8-item questionnaire designed to assess patient-reported cognitive deficits in individuals with MS. Each item is scored based on the frequency of cognitive difficulties experienced over the past month (0 = Never, 1 = Rarely, 2 = Sometimes, 3 = Fairly Often, 4 = Very Often). The scale includes four 2-item subscales-Executive/Speed, Working Memory, Expressive Language, and Episodic Memory-each with a total range of 0-8. A total score (range 0-32) is calculated by summing all item scores, with higher scores indicating greater cognitive impairment due to MS.
MIND Diet Score | Baseline, 6-months, and at 12-months
  Adherence to MIND Diet will be measured using MIND Diet score, where scores range 0-14. Higher scores indicate better adherence to a Mediterranean-style (MIND) diet and points are assigned based on how often an individual consumes the food group in question.
MIND Diet Adherence Score | Baseline, 6-months, and at 12-months
  Those assigned to the diet intervention arm will complete a self-assessment of their adherence to the MIND diet, indicating how closely an individual believes they are following the MIND diet. Scores range 0-100, where higher scores indicate greater diet adherence (100%=perfect adherence).
The Diet History Questionnaire (DHQ) | Baseline, 6-months, and at 12-months
  The Diet History Questionnaire (DHQ) is a 161-item survey measuring the frequency of specific food, beverage, and supplement intake. The DHQ is not scored; rather, it offers a detailed look into one's dietary patterns and nutrition by quantifying the nutrients, dietary constituents, and food groups that an individual has consumed over the past month.
The Insomnia Severity Index (ISI) | Baseline, 6-months, and at 12-months
  The Insomnia Severity Index (ISI) is a 7-item questionnaire designed to assess the severity of insomnia symptoms. Each item is scored from 0 to 4, with higher scores indicating more acute symptoms. The total score is calculated by summing the individual item scores, resulting in a total range of 0-28. Scores are categorized as follows: 0-7 (No clinically significant insomnia), 8-14 (Subthreshold insomnia), 15-21 (Clinical insomnia - moderate), and 22-28 (Clinical insomnia - severe).
The Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Baseline, 6-months, and at 12-months
  The Godin Leisure-Time Exercise Questionnaire (GLTEQ) is a tool used to assess weekly exercise habits, measuring both frequency (number of 15-minute sessions) and intensity (Light, Moderate, and Strenuous). A weekly leisure activity score is calculated using the formula: (9 × Strenuous) + (5 × Moderate) + (3 × Light). Higher scores indicate greater physical activity levels, with classifications as follows: ≥24 (Active), 14-23 (Moderately Active), and ≤14 (Insufficiently Active/Sedentary).
Glial fibrillary acidic protein (GFAP) level | Baseline, 6-months, and at 12-months
  GFAP is a protein expressed by astrocytes (supporting cells in the brain) that can be elevated in certain disorders like multiple sclerosis
Lipid panel | Baseline, 6-months, and at 12-months
  blood tests that measure the amount of fats in the blood
Apolipoproteins level | Baseline, 6-months, and at 12-months
  blood tests that measure the amount of fats in the blood
Hemoglobin A1C Test | Baseline, 6-months, and at 12-months
  A1C is a lab test that shows the average level of blood sugar (glucose) over the previous 3 months. It shows how well patients are controlling their blood sugar to help prevent complications from diabetes.
The NHANES biological aging index (BAI) | Baseline, 6-months, and at 12-months
  The NHANES Biological Aging Index (BAI) is a multi-marker index designed to estimate biological age relative to chronological age. It is derived from a mathematical equation that incorporates various biomarkers known to change with age. These biomarkers include resting blood pressure, forced expiratory volume (FEV1), and lab values such as serum creatinine, C-reactive protein, blood-urea nitrogen, albumin, alkaline phosphatase, cholesterol, cytomegalovirus (CMV) antibodies, and hemoglobin A1c. The index compares these values to a reference population of healthy individuals to estimate the rate of aging. A higher BAI score indicates faster aging of cells and tissues, while a lower score suggests slower aging. There is no defined minimum or maximum score for the BAI.
Leukocyte telomere length (LTL) | Baseline, 6-months, and at 12-months
  Leukocyte telomere length (LTL) measures biological aging (longer length associated with younger biological age). Biological age (BA) describes the extent of aging, based on the age of one's cells and tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana B Katz Sand, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared with qualified investigators upon request and review, in accordance with institutional policies.